CLINICAL TRIAL: NCT06969963
Title: Single-dose, Randomized, Two-period, Two-sequence Crossover Study to Evaluate the Bioequivalence of Lepsiramp 0.5mg/ml Oral Suspension (Test) and Fycompa® 0.5mg/ml Oral Suspension (Reference) Under Fasting Conditions
Brief Title: Bioequivalence Assessment Between Two Perampanel Oral Suspension Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aya Mohammed Abdel Magid Abdel Hamid (Other)
Collaborators: Advanced Research Center (ARC) (Unknown); Global Napi Pharmaceuticals for Global Advanced Pharmaceuticals (Unknown)
Responsible Party: Sponsor-Investigator, Aya Mohammed Abdel Magid Abdel Hamid, Lecturer of Clinical Pharmacy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE0124LEP0.5-GAP/01
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Bioequivalence Study in Healthy Subjects
Keywords: Perampanel; Bioequivalence; Oral suspension; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Suspensions; perampanel

STUDY DESIGN:
Intervention Model Description: single center, open label, randomized, single-dose, 2-sequence, 2-period, crossover, bioequivalence trial conducted under fasting conditions with healthy participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lepsiramp (perampanel 0.5 mg/mL) oral suspension (Active Comparator): Test Product
  Interventions: Drug: Lepsiramp, 0.5 Mg/mL Oral Suspension
- Fycompa® (perampanel 0.5 mg/mL) oral suspension (Active Comparator): Reference Product
  Interventions: Drug: Fycompa, 0.5 Mg/mL Oral Suspension

INTERVENTIONS:
Drug: Lepsiramp, 0.5 Mg/mL Oral Suspension — Test product
  Other Names: Perampanel 0.5mg/mL
  Arms: Lepsiramp (perampanel 0.5 mg/mL) oral suspension
Drug: Fycompa, 0.5 Mg/mL Oral Suspension — Reference product
  Other Names: perampanel 0.5mg/mL
  Arms: Fycompa® (perampanel 0.5 mg/mL) oral suspension

SUMMARY:
An open label, randomized, single-dose, two-sequences, two-periods, crossover study to assess the bioequivalence of perampanel in Lepsiramp 0.5mg/ml oral suspension (Test product) in comparison with Fycompa® 0.5mg/ml oral suspension (Reference product) in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
This was a single-dose, open-label, randomized, two-sequence, two-period crossover bioequivalence study conducted under fasting conditions at Advanced Research Center (ARC), Cairo, Egypt in 2024. The study compared the bioequivalence of Lepsiramp 0.5 mg/mL oral suspension (Test) with Fycompa® 0.5 mg/mL oral suspension (Reference), both formulations containing perampanel.

Study Design Participants were randomized in a 1:1 ratio to receive the test or reference product across two study periods, separated by a 6-week washout. Each subject received a single 24 mL oral dose (equivalent to 12 mg perampanel) under fasting conditions. A standardized diet was provided during each period, and fluid intake was controlled pre- and post-dosing to maintain consistency.

Blood Sampling Details In each period, 22 blood samples (5 mL each) were collected to characterize the plasma concentration-time profile. A forearm vein cannula was used for samples up to 24 hours; later samples were collected via venipuncture. Samples were centrifuged at 3500 rpm for 5 minutes at 4°C. Plasma was separated and stored at -80°C pending analysis.

Pharmacokinetic and Bioanalytical Methods Plasma perampanel concentrations were quantified using a validated LC-MS/MS method with a calibration range of 3-400 ng/mL. The primary PK parameters included Cmax and AUC₀-₇₂, while secondary parameters were Tmax, AUC₀-inf, t½, and ke. PK analysis was conducted using Phoenix WinNonlin (v8.3.4), with calculations based on actual sampling times.

Bioequivalence Evaluation Bioequivalence was determined if the 90% confidence intervals (CIs) for the geometric mean ratios (GMRs) of Cmax and AUC₀-₇₂ fell within the 80-125% range. ANOVA was applied to log-transformed data for Cmax and AUC, and Wilcoxon signed-rank test was used for Tmax comparisons.

Safety Evaluation Subjects were monitored for adverse events throughout the study. Vital signs were assessed at multiple time points (pre-dose, and 2, 6, 12, and 72 hours post-dose). Complete blood counts were performed at the study's end.

Statistical Analysis Sample size was calculated using R (v4.2.1), assuming a 19.35% intra-subject variability for Cmax, with 80% power, 5% significance level, and adjustment for expected dropouts. The Two One-Sided Tests (TOST) procedure was applied to log-transformed PK parameters to assess bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged between 18 and 55 years.
2. Non-smokers or mild smokers with a maximum limit of 5 cigarettes/day.
3. Normal physical examinations at screening visit.
4. Having BMI ranged between 18.5-30 kg/m2.
5. Ability to communicate adequately with the clinical staff.
6. Ability and agreement to comply with the study requirements.
7. Normal BP and HR measured under stabilized conditions.

   * The Blood pressure is considered normal if the SBP falls within 100 to 140 mmHg, and the DBP within 60 to 90 mmHg.
   * The heart rate normal range is from 60 to 100 bpm.
   * Respiratory rate normal range is from 12 to 16 breaths per minute.
   * Temperature normal range is from 36.5ºC to 37.5ºC.
8. Normal laboratory results within normal range or with clinically non-significant deviation including: Complete Blood Count, Clinical Chemistry: Random blood sugar, blood urea, creatinine, sodium, potassium, total bilirubin, alanine amino transferase (ALT/GPT), aspartate amino transferase (AST/GOT), alkaline phosphatase, total protein in serum, Lipid profile, urinalysis.
9. Negative Virology tests: HIV (HIV Ab), hepatitis B (HBsAg), hepatitis C (HCV IgG).
10. Negative results for abused drug analysis in urine (Amphetamine (AMP), Barbiturate (BAR), Benzodiazepine (BZO), Cannabinoid (THC), Cocaine, Opiates (Morphine (MOP), Tramadol (TRA)).
11. Understanding of the study and agreeing to give a written informed consent.
12. Using an adequate contraception method during the study and for at least 30 days after the study (for potential subjects).

Exclusion Criteria:

1. Subjects who have atopic constitution, asthma or known allergy for the API under investigation and/or any other ingredients of the investigational product.
2. Presence of clinical relevance of cardiovascular, neurological, musculoskeletal, hematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolism or psychiatric disease.
3. Symptomatic or asymptomatic orthostatic hypotension at screening defined by a decrease of SBP more than 20 mmHg or DBP more than 10 mmHg occurs between sitting/supine to standing position. The subject will be excluded (if the drug under investigation has antihypertensive properties or documented to have orthostatic hypotension as a side effect).
4. Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or herniotomy.
5. Subjects who have given more than 400 mL blood within the last two months before the first drug administration and subjects who have participated in any drug research within the last two months before the first day of drug administration.
6. Subjects who used any prescribed systemic medication (including OTC medication) within 2 weeks (or six elimination half-lives of this medication, whichever is longer) before the initiation of the study (except for single doses of analgesics which have no drug interaction with study product).
7. Use of any vitamins or herbal products within 3 days prior to the initial dose of the study medication.
8. Subjects who have any chronic disease which might interfere with the absorption, distribution, metabolism or excretion of the drug.
9. Subjects who consumed grapefruit or grapefruit juice during 48 hr prior to drug administration, during the study.
10. History of alcohol abuse and/or regular use of more than 2 units of alcohol per day or positive alcohol test.
11. History of difficulty of swallowing.
12. Intake of enzyme-inducing, organ toxic, long half-life drugs within 4 weeks before start of the study
13. Subjects who follow a special diet due to any reason, e.g., vegetarian.
14. Has a recent acute infection.
15. Pregnant females or female subjects who practice lactation or unprotected females with pregnancy potential

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Cmax | From time zero up to 72 hours in each study period
  Peak plasma concentration
AUC(0-72) | From time zero up to 72 hours in each study period
  The area under the plasma concentration-time curve up to 72 hours

SECONDARY OUTCOMES:
Tmax | From time zero up to 72 hours in each study period
  The time of the peak plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kamal A. Badr, Ph.D., Study Director — Advanced Research Center (ARC)
Locations (1):
- Advanced Research Center (ARC), Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] AbdelMagid AM, Badr KA, Rezk MR. Bioequivalence of Two Perampanel Oral Suspension Formulations in Healthy Subjects: A Randomized Crossover Study. Drugs R D. 2025 Dec;25(4):343-351. doi: 10.1007/s40268-025-00526-5. Epub 2025 Nov 18. PMID 41249688